CLINICAL TRIAL: NCT05509088
Title: Impact of the Early Use of High Flow Nasal Cannula in Patients With Post-traumatic Lung Contusion, a Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FAMSU R 116/ 2022
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Traumatic Lung Injury
MeSH Terms: conditions — Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high flow nasal cannula (Experimental): will receive oxygen through high flow nasal cannula
  Interventions: Device: high flow nasal cannula
- oxygen mask (No Intervention): will receive oxygen through oxygen mask

INTERVENTIONS:
Device: high flow nasal cannula — Patients in the intervention group receive oxygen through HFNC with a flow rate of set initially at 40 L / min, FiO2 adjusted to maintain SpO2 ≥ 92%, and will be humidified, heated to 34-37 °C, disconnection will be allowed only when ambulation is required, patients will be instructed to practice mouth closing throughout the HFNC therapy as much as possible
  Arms: high flow nasal cannula

SUMMARY:
We hypothesize that early and continuous administration of oxygen via high flow nasal cannula in patients with lung contusion and non-severe acute lung injury might reduce the incidence of intubation and hold the deterioration of pulmonary functions.

ELIGIBILITY:
Inclusion Criteria:

Willing and able to provide written informed consent prior to performing study procedures, currently hospitalized and requiring medical care for blunt chest trauma, within 24h of trauma

Exclusion Criteria:

* face trauma or surgery, airway obstruction, known to have chronic chest condition

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2022-12-28 (Estimated); Study Completion 2022-12-28 (Estimated)

PRIMARY OUTCOMES:
need for intubation and mechanical ventilation within 28 days of randomization. | 3 months
  the incidence of intubation in patients with lung contusion who receive oxygen through high flow nasal cannula

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No